CLINICAL TRIAL: NCT03689634
Title: Move For Surgery - A Novel Preconditioning Program to Optimize Health Before Thoracic Surgery: A Randomized Controlled Trial
Brief Title: Move For Surgery - A Novel Preconditioning Program
Acronym: MFS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other)
Responsible Party: Principal Investigator, Wael Hanna, Associate Professor of Surgery, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SJHH-MFS-RCT
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer, Nonsmall Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Move For Surgery Preconditioning Program Intervention Group (Experimental)
  Interventions: Device: Move For Surgery Preconditioning Program using a Wearable Activity Tracker (Fitbit) Intervention Group
- Standard Preoperative Care Group (No Intervention)

INTERVENTIONS:
Device: Move For Surgery Preconditioning Program using a Wearable Activity Tracker (Fitbit) Intervention Group — Participants randomized to this group will be be provided with a wearable activity tracker (Fitbit) for the duration of the study and asked to reach daily step goals.
  Arms: Move For Surgery Preconditioning Program Intervention Group

SUMMARY:
Lung cancer is the leading cause of cancer death in Canada. Most patients with this cancer will undergo treatment with major chest surgery that is associated with serious complications. As many as 50% of patients will suffer respiratory complications after surgery, keeping them in the hospital for extended periods of time. These long hospitalizations have a dramatic negative effect on the lives of those people, in addition to a large cost burden on our healthcare system. Traditionally, patients who suffer from complications are treated with rehabilitation AFTER the complications have occurred. But what if complications can be prevented BEFORE they happen? Having major chest surgery imposes great stress on the human body, one that is equivalent to running a marathon. Analogous to training before completing a marathon, the investigator designed Move For Surgery (MFS), a novel preconditioning program that encourages and empowers patients to improve their health prior to surgery. The investigator aims to demonstrate that patients who train with Move For Surgery will have lower respiratory complication rates, will recover better, and will leave the hospital sooner than their counterparts.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical stage I, II, or IIIa non-small cell lung cancer (NSCLC)
* Candidates for thoracic surgery, as determined by the operating surgeon

Exclusion Criteria:

* Clinical stage IIIb or IV NSCLC
* Patients with affected mobility (wheelchair, walker)
* Patients who use oxygen at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the comparative trial will be length of stay (LOS) in hospital after surgery, which will also be used to measure speed of recovery from surgery and postoperative complications. | 24 months
  LOS is a good surrogate measure for the speed of recovery from surgery (patients who recover faster leave hospital earlier) and postoperative complications (patients who do not suffer complications leave the hospital earlier).

SECONDARY OUTCOMES:
Secondary outcome will include differences in the 36-Item Short Form Health Survey (SF-36) scores before and after the intervention. | 24 months
  The quality of life as reported by patients will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Patel YS, Sullivan KA, Churchill IF, Beauchamp MK, Wald J, Mbuagbaw L, Fahim C, Hanna WC. Preconditioning program reduces the incidence of prolonged hospital stay after lung cancer surgery: Results from the Move For Surgery randomized clinical trial. Br J Surg. 2023 Oct 10;110(11):1467-1472. doi: 10.1093/bjs/znad252. PMID 37643916